CLINICAL TRIAL: NCT03022682
Title: Development of a Multi-Ethnic, Multimodal Obesity Cohort
Brief Title: Inflammation, Diabetes, Ethnicity and Obesity Cohort
Acronym: IDEO
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 14-14248
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Diabetes Mellitus; Pre Diabetes
Keywords: ethnicity; inflammation; obesity; diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Glucose Intolerance; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, Adipose tissue, stool

GROUPS / COHORTS (1):
- IDEO Cohort: Adipose tissue samples are collected from all participants, including aspirational subcutaneous biopsies from nonsurgical participants and excisional biopsies, performed intra-operatively by surgical collaborators as required.
  Participants also undergo anthropometric measurements, stool collection, blood sample collection for circulating blood cells, serum, and plasma.
  Dual-energy x-ray absorptiometry (DXA) scan for amount and distribution of body fat as well as bone density is performed.
  Study participants complete validated questionnaire inventories to measure bio-behavioral issues such as depression, stress, health locus of control, and dietary habits.

SUMMARY:
Obesity affects over one third of US adults (>72 million, with BMI ≥30 kg/m2), and the proportion of US adults with BMI ≥40 kg/m2 has doubled in the last 20 years. Obesity is associated with increased mortality through its linkage to comorbidities including diabetes, hypertension, dyslipidemia, osteoarthritis, sleep apnea and psychosocial disturbances. Given its prevalence, impact on morbidity and mortality, and economic cost, limiting the spread of obesity and its consequences is one of the most important problems of our time.

In this proposed study, investigators will recruit participants from a wide range of body mass index (BMI), ethnicity and Diabetes risk to collect data and blood, stool and adipose tissue samples in the San Francisco bay area.

DETAILED DESCRIPTION:
The Inflammation, Diabetes, Ethnicity and Obesity (IDEO) cohort is recruiting 350 individuals from various ethnicities, covering a spectrum of weight and Diabetes risk. The study is looking for participants between the ages of 18-75 years that are healthy with or without diabetes with a stable weight. The study will also like to include people who are slated to undergo any type of bariatric surgery for obesity or any other type of abdominal surgery at UCSF.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be healthy individuals between the ages of 18-75 years. These cutoffs are designed to allow inclusion of postmenopausal women, and younger/more active patients who are increasingly undergoing bariatric surgery.
* Patients with either diabetes type 2 or the metabolic syndrome will be included in the cohort.

Exclusion Criteria:

* Participants with chronic kidney disease (> stage 4)
* Autoimmune/inflammatory disease (e.g., Lupus, Ulcerative Colitis, etc.)
* Unstable angina, New York (NY) class III or IV congestive heart failure or myocardial infarction within 3 months of entry
* Clinically significant liver disease (e.g. Cirrhosis or liver failure)
* Weight > 450 pounds (DXA scan weight limit)
* History of organ transplant
* Treatment with chemotherapy or radiation therapy at the time of enrollment in study.
* Poorly controlled asthma (participants requiring inhaled glucocorticoids and/or oral glucocorticoids)
* Current nasal corticosteroid use (within the past month)
* Excessive alcohol or substance abuse
* Current use of anabolic steroids or testosterone for bodybuilding purposes. Testosterone use is permitted if prescribed for hypogonadism and dose stable for the past 6 months.
* Patients actively enrolled in interventional trials involving investigational agents
* Pregnant or breast-feeding women
* Appears unlikely or unable to participate in the required study procedures as assessed by the investigator, study coordinator or designee.
* History of abnormal clotting
* Previous bariatric surgery
* Anticoagulant use
* Methadone medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: IDEO Cohort participants
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2015-02; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Complete recruitment of IDEO cohort participants to spur novel and creative interactions between investigators that have transformative potential in obesity research. | 7 years
  Number of biological samples collected

SECONDARY OUTCOMES:
Adipose tissue inflammation and fibrosis | 7 years
  Quantification of pro-fibrotic and pro-inflammatory markers in the visceral and subcutaneous adipose tissue

CONTACTS AND LOCATIONS:
Overall Officials: Suneil Koliwad, MD,PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Koppel N, Bisanz JE, Pandelia ME, Turnbaugh PJ, Balskus EP. Discovery and characterization of a prevalent human gut bacterial enzyme sufficient for the inactivation of a family of plant toxins. Elife. 2018 May 15;7:e33953. doi: 10.7554/eLife.33953. PMID 29761785